CLINICAL TRIAL: NCT04235712
Title: Implementation of Harmonized Depression Outcome Measures in a Health System to Support Patient-Centered Outcomes Research
Brief Title: Implementation of Harmonized Depression Outcome Measures in a Health System
Status: Completed | Type: Observational
Sponsor: OM1, Inc. (Industry)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AHRQ_DEP_Health_System
Record Dates: First submitted 2020-01-07; First posted 2020-01-22 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Major Depression; Dysthymia
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Harmonized Depression Outcome Measures — This is an observational study where outcome measures will be extracted from patients' medical records and from questionnaires to provide information back to the clinician.

SUMMARY:
Working with a health system, the investigators will recruit practices to participate in the pilot study, consent and enroll patients with major depressive disorder, and collect the PHQ-9 from those patients at three timepoints (baseline, 6 months post-enrollment, and 12 months post-enrollment). The PHQ-9 will be captured either at an office visit or directly from patients. The investigators will build and implement an open-source SMART on FHIR app to collect key data from the EHR, combine that data with the PHQ-9 results, and present the measurements back to the clinicians. The investigators will then obtain feedback from clinicians on the value and usefulness of the app.

DETAILED DESCRIPTION:
The study is a longitudinal, observational pilot study that will assess the utility and value displaying the harmonized outcomes data to clinicians in the clinical workflow using an open-source, SMART on FHIR app. The app will connect with the site EHR, aggregate EHR and PRO data, calculate the outcome measure results, and return the results to the EHR so that they are viewable within the clinician workflow. Baseline data on patient characteristics, treatments, and symptoms will be combined with longitudinal data on outcomes during the study timeframe. All data will be collected from institution electronic medical records (EMRs), PRO portals, and other existing data sources, as needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* Diagnosis of major depression or dysthymia
* Willing and able to provide informed consent

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will collect data on approximately 50 patients with a diagnosis of major depression or dysthymia from a total of five practices within the same health system.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Death from suicide | 12-month intervals
  Patient age 18 or older with a diagnosis of major depression or dysthymia who died from suicide, reported in 12-month intervals.
Improvement in Depressive Symptoms: Remission | Baseline
  Patient Health Questionnaire-9 score > 9 who demonstrates remission defined as a Patient Health Questionnaire-9 score less than 5. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Improvement in Depressive Symptoms: Remission | 6 months post baseline (+/- 60 days)
  Patient Health Questionnaire-9 score > 9 who demonstrates remission defined as a Patient Health Questionnaire-9 score less than 5. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Improvement in Depressive Symptoms: Remission | 12 months post baseline (+/- 60 days)
  Patient Health Questionnaire-9 score > 9 who demonstrates remission defined as a Patient Health Questionnaire-9 score less than 5. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Improvement in Depressive Symptoms: Response | Baseline
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 score > 9 who demonstrates a response to treatment defined as a Patient Health Questionnaire-9 score that is reduced by 50% or greater from the initial Patient Health Questionnaire-9 score. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Improvement in Depressive Symptoms: Response | 6 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 score > 9 who demonstrates a response to treatment defined as a Patient Health Questionnaire-9 score that is reduced by 50% or greater from the initial Patient Health Questionnaire-9 score. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Improvement in Depressive Symptoms: Response | 12 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 score > 9 who demonstrates a response to treatment defined as a Patient Health Questionnaire-9 score that is reduced by 50% or greater from the initial Patient Health Questionnaire-9 score. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Worsening in Depressive Symptoms: Recurrence | Baseline
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 > 9 who demonstrates remission (defined as a Patient Health Questionnaire-9 score < 5) of at least two months' duration and subsequently experiences a recurrence of a depressive episode, defined as a Patient Health Questionnaire-9 score > 9 OR hospitalization for depression or suicidality. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Worsening in Depressive Symptoms: Recurrence | 6 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 > 9 who demonstrates remission (defined as a Patient Health Questionnaire-9 score < 5) of at least two months' duration and subsequently experiences a recurrence of a depressive episode, defined as a Patient Health Questionnaire-9 score > 9 OR hospitalization for depression or suicidality. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Worsening in Depressive Symptoms: Recurrence | 12 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 > 9 who demonstrates remission (defined as a Patient Health Questionnaire-9 score < 5) of at least two months' duration and subsequently experiences a recurrence of a depressive episode, defined as a Patient Health Questionnaire-9 score > 9 OR hospitalization for depression or suicidality. Patient Health Questionnaire scores range from 0 to 27. A higher score means more severe depression.
Adverse Events | Baseline
  Depression treatment-related adverse events, captured using the Frequency, Intensity, and Burden of Side Effects Ratings scale where available and extracted from data routinely recorded in the Electronic Medical Record. The Frequency, Intensity, and Burden of Side Effects Ratings score ranges from 0 to 6. A higher score means more of a burden.
Adverse Events | 6 months post baseline (+/- 60 days)
  Depression treatment-related adverse events, captured using the Frequency, Intensity, and Burden of Side Effects Ratings scale where available and extracted from data routinely recorded in the Electronic Medical Record. The Frequency, Intensity, and Burden of Side Effects Ratings score ranges from 0 to 6. A higher score means more of a burden.
Adverse Events | 12 months post baseline (+/- 60 days)
  Depression treatment-related adverse events, captured using the Frequency, Intensity, and Burden of Side Effects Ratings scale where available and extracted from data routinely recorded in the Electronic Medical Record. The Frequency, Intensity, and Burden of Side Effects Ratings score ranges from 0 to 6. A higher score means more of a burden.
Suicide Ideation and Behavior | Baseline
  Selection of 'several days', 'more than half the days' or 'nearly every day' option on Patient Health Questionnaire-9 item 9 ("Thoughts that you would be better off dead or of hurting yourself in some way") and/or documentation of nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, or active suicidal ideation extracted from data routinely recorded in the Electronic Medical Record. A higher score means more severe depression.
Suicide Ideation and Behavior | 6 months post baseline (+/- 60 days)
  Selection of 'several days', 'more than half the days' or 'nearly every day' option on Patient Health Questionnaire-9 item 9 ("Thoughts that you would be better off dead or of hurting yourself in some way") and/or documentation of nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, or active suicidal ideation extracted from data routinely recorded in the Electronic Medical Record. A higher score means more severe depression.
Suicide Ideation and Behavior | 12 months post baseline (+/- 60 days)
  Selection of 'several days', 'more than half the days' or 'nearly every day' option on Patient Health Questionnaire-9 item 9 ("Thoughts that you would be better off dead or of hurting yourself in some way") and/or documentation of nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, or active suicidal ideation extracted from data routinely recorded in the Electronic Medical Record. A higher score means more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Baystate Health, Springfield, Massachusetts, United States

REFERENCES:
- See also: AHRQ webpage containing details on this initiative — https://effectivehealthcare.ahrq.gov/products/registry-of-patient-registries/outcome-measure-harmonization

DOCUMENTS (1):
  • Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04235712/ICF_000.pdf